CLINICAL TRIAL: NCT01703728
Title: SHOview Observational Study. Controlled Ovarian Stimulation by HP-hMG for IVF / ICSI Cycles: Study on Ovarian Hyper Stimulation Syndrome in a Cohort of Women From 18 to 36 Years Old.
Brief Title: Controlled Ovarian Stimulation by HP-hMG for IVF / ICSI Cycles: Study on Ovarian Hyper Stimulation Syndrome in a Cohort of Women From 18 to 36 Years Old.
Acronym: SHOview
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000012
Record Dates: First submitted 2012-10-03; First posted 2012-10-10 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Ovarian Hyperstimulation Syndrome (OHSS)
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — No biological samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Highly purified menotropin (HP-hMG) treatment: Cohort of women from 18 to 36 years old treated by HP-hMG for controlled ovarian stimulation (COS) for a first or second cycle of IVF / ICSI.
  Interventions: Other: Highly purified menotropin (HP- hMG) treatment

INTERVENTIONS:
Other: Highly purified menotropin (HP- hMG) treatment — No intervention: patients treated by highly purified menotropin for COS according to physicians' current practice

SUMMARY:
Ovarian hyper stimulation syndrome (OHSS) is a potentially serious complication of ovarian stimulation in IVF (In Vitro Fertilisation). The main objective of this study is to describe the incidence of moderate or severe forms of OHSS in women between 18 and 36 years of age treated with HP-hMG.

ELIGIBILITY:
Inclusion Criteria:

* Women who present infertility of more than one year and are candidates for a first or second IVF cycle with or without ICSI for whom HP-hMG is prescribed for COS.
* Absence of infertility treatment during the last 3 months before enrolment.
* Age: from 18 to 36 years old.
* BMI between 18 and 30 kg / m².
* Presence of both ovaries accessible to puncture and absence of ovarian or uterine abnormalities.
* Male or female infertility.
* Ovarian stimulation by HP-hMG with pituitary desensitization by a GnRH agonist or antagonist.
* Normal ovarian reserve according to physician habitual evaluation.
* Consent to participate of the no-interventional study and signature of the patients' information sheet.

Exclusion Criteria:

* Presence of a chronic disease, cancer or endocrine disease that could potentially influence the results of the stimulation or that represents a contraindication for ovarian stimulation.
* Known endometriosis grade III or IV.
* Contraindication to the use of gonadotropins or current pregnancy diagnosed by the clinician.
* Recurrent miscarriages, known genetic disease of one of the partners or indication of a preimplantation genetic diagnosis (PGD).
* Smoking over than 10 cigarettes / day.´
* Participation in an interventional study at the time of inclusion.
* Known poor ovarian response in a previous cycle of stimulation (number of oocyte collected ≤ 3, and / or more than 2 previous IVF/ICSI cycles and / or abnormal result in ovarian reserve test (AMH < 1 ng/ml with Immunotech equipment or AMH<0.7 ng/ml with DSL equipment).

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women from 18 to 36 years old treated by HP-hMG for controlled ovarian stimulation (COS) for a first or second cycle of IVF / ICSI.
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Incidence of moderate/severe OHSS | 2-12 weeks

SECONDARY OUTCOMES:
Incidence of each form of OHSS: mild, moderate and severe | 2-13 weeks
Incidence of moderate and of severe OHSS among patients treated by a GnRH agonist or antagonist desensitization protocol | 2-13 weeks
OHSS clinical features description according to the Royal College of Obstetricians and Gynaecologists classification | 2-13 weeks
Patients' baseline characteristics | At baseline
Dosage adjustment, modification of the treatment, coasting and cycle cancellation, no hCG administration and embryo transfer cancellation | Up to 3 weeks
Description and duration of hospitalisation, treatments prescribed | 2-13 weeks
Frequency and reasons for stimulation arrest and no embryo transfer decision | 2-4 weeks
Number of oocytes retrieved, number of mature oocytes, fertilization rate, embryo quality, embryo freezing, number and quality of transferred embryos | 2-3 weeks
Description of serious and not serious adverse events | 2-13 weeks
Description of patient's compliance to the prescribed treatment | 2-4 weeks
Clinical pregnancy rate, spontaneous miscarriage and ongoing pregnancy rate | 4-13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (20):
- France (20):
  - Cabinet Mirabeau Roy René (there may be other sites in this country), Aix-en-Provence
  - Hôtel Dieu, Angers
  - Clinique La Chataigneraie, Beaumont
  - CHU Pellegrin, Bordeaux
  - Clinique Léonard de Vinci, Chambray-lès-Tours
  - CHI, Créteil
  - Hôpital Victor Jousselin, Dreux
  - Institut Rhonalpin, Écully
  - Cabinet Médical Maréchal Leclerc, Grenoble
  - Groupe Hospitalier du Havre - Hôpital Jacques Monod, Le Havre
  - Cabinet Médical Lille avenue de Dunkerque, Lille
  - Hôpital Jeanne de Flandre, Lille
  - Hôpital Privé Natecia, Lyon
  - CHU de Marseille -Hôpital Conception, Marseille
  - Hôpital Maternité de Metz, Metz
  - CHU de Nantes, Nantes
  - Cabinet Médical de Prony, Paris
  - Hôpital St Vincent de Paul, Paris
  - CHU de Rennes, Rennes
  - Clinique Mutualiste La Sagesse, Rennes

REFERENCES:
- [Result] Barriere P, Dewailly D, Duhamel A, Gayet V. [Ovarian hyperstimulation syndrome after stimulation with highly purified hMGfor in vitro fertilization: Observational study SHOview]. Gynecol Obstet Fertil Senol. 2017 May;45(5):283-290. doi: 10.1016/j.gofs.2017.03.004. Epub 2017 Apr 29. French. PMID 28461237